CLINICAL TRIAL: NCT06418139
Title: Etude de l'Effet de l'Horaire de Perfusion de l'immunothérapie Sur la réponse et la toxicité Des Traitements Chez Les Patientes Atteintes de Cancer du Sein Triple négatif à Haut Risque traité Par chimiothérapie néoadjuvante et Pembrolizumab
Brief Title: Association of Pembrolizumab Infusion Time and Efficacy in Patients With Non-metastatic Triple-negative Breast Cancer (TNBC) Treated With Neoadjuvant Chemotherapy and Immunotherapy
Acronym: PEMCLOCK
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240393
Record Dates: First submitted 2024-04-19; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Non-Metastatic Breast Carcinoma
Keywords: Non metastatic Triple-negative breast cancer; Triple-negative breast cancer; Chronotherapy; Immunotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Morning group
  Interventions: Other: No intervention
- Afternoon group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention added by the study

SUMMARY:
Background: Triple negative breast cancer (TNBC) is characterized by an aggressive biological behaviour responsible for higher risk of recurrence and shorter median survival. Pembrolizumab, an immune checkpoint inhibitor (ICI) targeting programmed death (PD-1), in association to chemotherapy showed improvement of event-free survival in patients with previously untreated stage II or III TNBC and has been approved in Europe since March 2022 for this indication (KEYNOTE-522). Circadian timing system controls many various biological functions in humans including xenobiotic metabolism and elimination, immune functions, cell cycle event and apoptosis. Thus, chronotherapeutic approaches have shown improved efficacy and tolerability in the treatment of different types of cancer, notably in colorectal cancer. Pronounced circadian rhythms in immune functions are generated by cell-autonomous molecular clocks in T and B lymphocytes, macrophages, neutrophils, and dendritic cells. Recently, first evidence of the effect of timing infusion of immune checkpoint inhibitors on prognosis of patients with cancer has been reported in several retrospective trials. Landre et al.'s meta-analysis of 7 retrospective studies including 1019 patients who had metastatic cancer was presented at the American Society of Clinical Oncology (ASCO) meeting in 2023. An early time-of-day ICI infusions was associated with an increase overall survival (HR: 0.49, [95% CI: 0.36-0.69] p < 0.0001).

Objectives: The aim is to analyze immunotherapy infusion timing impact on histological response, toxicity and Event Free-Survival (EFS) in patients with TNBC treated with Neo-Adjuvant Chemotherapy (NAC) associated with pembroluzimab. Measure of histological response is the primary objective determined by Residual Cancer Burden (RCB). Secondary endpoints are Event free Survival (EFS), calculated from the date of diagnosis to invasive local, regional, or metastatic relapse, contralateral breast cancer, or death from any cause), toxicity which is assessed by recording adverse events (CT-CAE v5) occurring from start of treatment to last course.

Methods: Data from patients with histologically proven early TNBC treated from July 2021 to May 2023 with the association of Pembrolizumab, Paclitaxel Carboplatine followed with Pembrolizumab Cyclophosphamide Epirubicine (according to KEYNOTE 522 study) will be collected. Dosing times of each Pembrolizumab and chemotherapy infusions given to consecutive patients as a neoadjuvant standard treatment, associated with chemotherapy, for early TNBC are retrieved from hospital records. Adjuvant Pembrolizumab timing intake will be also recorded as EFS is a secondary endpoint.

Statistics: First, median clock hour of all infusions of Pembrolizumab will be determined. Then, patients will be dichotomized between "morning' and 'afternoon' groups using 2 cut-offs: 1/ median clock of all infusions of pembrolizumab ('morning group' will include the patients who receive the majority of Pembrolizumab infusions before this median clock hour and 'afternoon group', patients who receive the majority of Pembrolizumab infusions after this median clock hour) and 2/ cut-off optimizing differences of RCB between two groups.

Patient's characteristics, toxicities, tumor response and EFS will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age ≥ 18 years-old
* Previously untreated histologically proven triple-negative breast cancer (RE < 10%, RP < 10%, Her-2 negative)
* No metastatic
* Having at least one injection of pembrolizumab associated with chemotherapy
* Pembrolizumab injection schedule correctly reported by the nurse in charge of the patient

Exclusion Criteria:

• Metastatic disease

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female with high-risk early triple-negative breast cancer treated with neoadjuvant chemotherapy combined with pembrolizumab
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Residual cancer burden class (RCB) | Up to 36 months
  RCB is studied after neoadjuvant treatment (Symmans et al. 2007)

SECONDARY OUTCOMES:
Number of immune adverse events | Up to 36 months
  Measurement of immune adverse events according to CTC-CAE Toxicity Grading Scale for Determining The Severity of Adverse Events version 5
Histological Complete Response (hCR) rate versus invasive residual disease rate | Up to 36 months
  Complete response is defined as hCR or RCB 0 Invasive residual disease rate is defined as RCB 2-3
Tumor-infiltrating lymphocyte (TIL) levels | Up to 36 months
  Association of RCB (class and continuous variable) with tumor-infiltrating lymphocyte (TIL) levels
Progression-free survival | At 2 years
Number of Pembrolizumab infusions performed | Up to 36 months
Tumor cellularity | Up to 36 months
  in %
Size of residual breast tumor | Up to 36 months
  mm x mm
Number of invaded nodes | Up to 36 months
Diameter of largest lymph node metastasis if lymph node invaded | Up to 36 months